CLINICAL TRIAL: NCT00938834
Title: A Randomized Controlled Trial Of Qigong For Treatment Of Fibromyalgia
Brief Title: Qigong For Treatment Of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Mary Lynch, MD FRCPC, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RS/2010-094
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Fibromyalgia Pain

ARMS (1):
- CFQ Qigong training group (Active Comparator): Qigong training con- sisted of an initial workshop conducted over three con- secutive half-days by a qualified CFQ instructor. Participants received training in level 1 CFQ; this con- sisted of instruction in seven key movements known as "the hexagram" and ancillary exercises. Hexagram move- ments consist of choreographed movements that emphasize softness, relaxation, downward releases and full body distribution of "qi". Once initial training was complete, participants were asked to practice CFQ at home for 45 to 60 minutes per day for eight weeks; time could be broken up into shorter sessions during the day. Participants returned for a 60 minute weekly review/group practice sessions for these eight weeks.
  Interventions: Other: CFQ Qigong

INTERVENTIONS:
Other: CFQ Qigong — CFQ Qigong training session training will consist of three half days of training in the technique. Following the training sessions, participants will return to the study site on a weekly basis for the first 8 weeks.

SUMMARY:
Fibromyalgia is a syndrome characterized by widespread musculoskeletal pain and hyperalgesia with a prevalence of 2-4% in the general population; it is often accompanied by fatigue, insomnia, anxiety, depression and other conditions. It is a difficult condition to treat, and only recently have drugs been approved by the FDA specifically for the treatment of this condition (Lyrica was approved in 2007, Duloxetine in 2008). There are now several clinical trials of drugs commonly used to treat neuropathic pain (amitriptyline, gabapentin, pregabalin, acetaminophen/tramadol, duloxetine, minserin) reporting some degree of efficacy in treating fibromyalgia. This efficacy makes it practical to consider fibromyalgia along with other neuropathic pain conditions. However, such drug trials report only partial efficacy in relieving pain and/or other symptoms. Current treatment recommendations indicate the need for a multimodal approach; this includes medical management using appropriate drug therapies, psychological therapies, exercise and complementary approaches. The current proposal is for a randomized controlled trial to compare qigong (a complementary modality) to a wait list control to determine if qigong is a useful complementary therapy for fibromyalgia.

The investigators recently completed a pilot trial in which they examined a specific form of qigong (CFQ Qigong, available locally in Halifax), and observed beneficial effects against pain, fibromyalgia impact, and on quality of life scores; importantly, these benefits were all sustained for 6 months to the end of the trial. On the basis of these preliminary observations, the investigators now propose a controlled trial in which CFQ Qigong is compared to a wait list control group. The latter group will be offered qigong training at the end of the trial, so could really be characterized as a delayed treatment group. The study will consist of a 3-day training period, weekly review of technique sessions for 8 weeks, daily practice for 8 weeks, with assessments at baseline, at 8 weeks following the training and practice, and follow-up assessments at 4 and 6 months. Study outcomes will include: (a) pain (numeric rating scale - pain intensity), (b) impact (fibromyalgia impact questionnaire), (c) quality of life measures (SF-36), (d) patient assessments (patient global impression of change and satisfaction scales), (e) sleep measures (Pittsburgh sleep quality index, actigraphy, sleep diary). In addition to these assessments, the investigators will also conduct qualitative assessments in which participants provide a more open-ended assessment of their health status at these same intervals. The main hypothesis being examined is that CFQ Qigong will produce benefits compared to the wait list group.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* A diagnosis of fibromyalgia according to American College of Rheumatology criteria
* Moderate to severe pain, as defined by an average 7-day pain score of greater than 4.0 on an 11-point numerical rating scale for pain intensity
* Pain medications must have been stable for at least 14 days.
* Ability to follow the protocol (with reference to cognitive and situational conditions, (e.g. stable housing, ability to attend follow-up visits, motivation and commitment to self practice of CFQ Qigong for 45-60 minutes per day).
* Willing and able to give written informed consent

Exclusion Criteria:

* Presence of clinically significant medical disorder on history or physical exam that would compromise the participants' safety in the trial as judged by the study physician
* Already practicing CFQ Qigong on a regular basis
* Unable to commit to 45-60 minutes of CFQ Qigong practice per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the change in mean daily pain diary score from baseline (average pain score over 7 days pre-treatment) to the final week of Qigong treatment. | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Management Unit - CDHA, Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Lynch M, Sawynok J, Hiew C, Marcon D. A randomized controlled trial of qigong for fibromyalgia. Arthritis Res Ther. 2012 Aug 3;14(4):R178. doi: 10.1186/ar3931. PMID 22863206
- [Derived] Castro MP, Goldstein N. Mismatch repair deficiency associated with complete remission to combination programmed cell death ligand immune therapy in a patient with sporadic urothelial carcinoma: immunotheranostic considerations. J Immunother Cancer. 2015 Dec 15;3:58. doi: 10.1186/s40425-015-0104-y. eCollection 2015. PMID 26674132